CLINICAL TRIAL: NCT00895739
Title: Alemtuzumab and Low-Dose Cyclosporine-A as Alternative Immunosuppressive Treatment for Severe Aplastic Anemia (SAA) and Single-Lineage Aplastic Patients
Brief Title: Alemtuzumab and Low-Dose Cyclosporine in Treating Patients With Severe Aplastic Anemia or Acquired Marrow Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: UNMS-ALESAA; CDR0000639649 (Registry Identifier: PDQ (Physician Data Query)); EU-20927; EUDRACT-2008-001151-22
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-05

CONDITIONS: Nonmalignant Neoplasm
Keywords: aplastic anemia
MeSH Terms: conditions — Neoplasms; Anemia, Aplastic | interventions — Alemtuzumab; Cyclosporine

INTERVENTIONS:
Biological: alemtuzumab
Drug: cyclosporine

SUMMARY:
RATIONALE: Immunosuppressive therapies, such as alemtuzumab and cyclosporine, may improve bone marrow function and increase blood cell counts. Giving alemtuzumab together with cyclosporine may be an effective treatment for severe aplastic anemia or acquired marrow failure.

PURPOSE: This phase II trial is studying the side effects of giving alemtuzumab together with cyclosporine and to see how well it works in treating patients with severe aplastic anemia or acquired marrow failure.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of alemtuzumab and low-dose cyclosporine, as defined by occurrence of adverse effects, in patients with severe aplastic anemia or single lineage acquired marrow failure.
* Determine the efficacy of this regimen, in terms of overall survival, hematological response (partial and complete response, including time to response) and failure-free survival (failure is defined as no response, chronic treatment-maintained response, or relapse), in these patients.

Secondary

* Evaluate the incidence of adverse effects after treatment.
* Evaluate the long-term safety of alemtuzumab treatment.
* Determine the time to achieve a complete hematological response.
* Determine the proportion of patients maintaining hematological response free of any treatment.
* Determine the incidence of relapse in responding patients.
* Determine the incidence of severe infections.
* Determine the requirement for IV antibiotics and antifungal therapy.
* Determine the requirement for red cell and platelet transfusion.
* Determine the incidence of CMV reactivation.
* Determine the kinetics of immune reconstitution.
* Determine the incidence of paroxysmal nocturnal hemoglobinuria clone (lymphoid or myeloid) development.
* Determine the incidence of clonal evolution (i.e., karyotypic abnormalities or secondary myelodysplasia/leukemia).

OUTLINE: Patients receive alemtuzumab subcutaneously on days 1-5*. Patients also receive oral cyclosporine beginning on day 7 and continuing for ≥ 180 days, followed by a taper according to clinical condition.

NOTE: *Patients with single lineage aquired marrow failure receive alemtuzumab on days 1-4.

After completion of study therapy, patients will be followed up every 3 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Severe or very severe aplastic anemia, as defined by the following criteria:

    * Meets ≥ 2 of the following criteria:

      * Absolute neutrophil count < 0.5 x 10^9/L (severe) or < 0.2 x 10^9/L (very severe)
      * Platelet count < 20 x 10^9/L
      * Reticulocyte count < 20 x 10^9/L
    * Hypocellular bone marrow (< 30% cellularity) without evidence of fibrosis or malignant cells
  * Single lineage acquired marrow failure (e.g., pure red cell aplasia, agranulocytosis, amegakaryocytic thrombocytopenia)
* Paroxysmal nocturnal hemoglobinuria clone allowed
* Failed first-line therapy with antithymocyte globulin (ATG) and cyclosporine OR not eligible for ATG-based studies

  * Failure is defined as lack of hematological response, requirement for chronic immunosuppressive treatment to sustain response, or relapse
* Not eligible for a low-risk stem cell transplantation
* No evidence of risky myelodysplastic syndromes (i.e., IPSS 3-4), as defined by the presence of marrow blast excess or karyotypic abnormalities, or other primitive marrow disease
* No history of constitutional aplastic anemia (e.g., Fanconi anemia or dyskeratosis congenita)

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Not pregnant or nursing
* No active malignant tumor within the past 5 years
* Transaminases ≤ 3 times upper limit of normal (ULN)
* Albumin ≥ 1.5 g/L
* Creatinine ≤ 3 times ULN
* No CMV viremia, as defined by positive PCR or pp65 test
* No cardiac failure (i.e., ejection fraction < 35%)
* No other concurrent life-threatening disease (including HIV infection)

PRIOR CONCURRENT THERAPY:

* No prior allogeneic stem cell transplantation
* At least 2 weeks since prior cyclosporine or filgrastim (G-CSF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Safety, as defined by occurrence of adverse effects
Overall survival
Hematologic response (partial and complete response, including time to response)
Failure-free survival (failure is defined as no response, chronic treatment-maintained response, or relapse)

SECONDARY OUTCOMES:
Incidence of adverse effects after treatment
Long-term safety of alemtuzumab treatment
Time to achieve a complete hematological response
Proportion of patients maintaining hematological response free of any treatment
Incidence of relapse in responding patients
Incidence of severe infections
Requirement for IV antibiotics and antifungal therapy
Requirement for red cell and platelet transfusion
Incidence of CMV reactivation
Kinetics of immune reconstitution
Incidence of paroxysmal nocturnal hemoglobinuria (PNH) clone (lymphoid or myeloid) development
Incidence of clonal evolution (i.e., karyotypic abnormalities or secondary myelodysplasia/leukemia)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Rotoli, MD, Principal Investigator — Federico II University
Locations (1):
- Federico II University Medical School, Naples, Italy